CLINICAL TRIAL: NCT05175976
Title: Patient Safety in the Operating Room: Helsinki Declaration Implementation in Ukraine
Status: Completed | Type: Observational
Sponsor: Bogomolets National Medical University (Other)
Responsible Party: Principal Investigator, Kateryna Bielka, Assistant professor at the Department of OF SURGERY, ANESTHESIOLOGY AND INTENSIVE THERAPY OF POSTGRADUATE EDUCATION, Bogomolets National Medical University
Other Study IDs: K44YB21yi7
Record Dates: First submitted 2021-11-30; First posted 2022-01-04 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Safety Issues
Keywords: patient safety; monitoring; Helsinki Declaration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Athe study to evaluate the implementation of the components of the Declaration of Helsinki in Ukrainian hospitals, as well as other safety measures during surgeries.

DETAILED DESCRIPTION:
A study was conducted from May 2021 to September 2021 at the Ukrainian hospitals. The study design was approved by the Ethical Committee at Bogomolets National Medical University. The survey was conducted by filling out a standard Google form. The link to the survey was distributed on the official page of the Association of Anesthesiologists of Ukraine, through social networks Facebook and Instagram on the official webpages of the Department of Surgery, Anesthesiology and Intensive Care of the Institute of Postgraduate Education of NMU. O.O. Worshipers. A total of 174 respondents took part in the survey.

To conduct the survey, we formed a questionnaire of 24 items. The questionnaire was designed to ensure sufficient collection of data from respondents on demographics, awareness of the Declaration, and the use in the everyday practice of the measures recommended in it to promote patient safety. However, the structure of the questionnaire allowed people to fill it in a short time. We also provided respondents with more descriptive and detailed answers to some questions if they wished. The survey was conducted in Ukrainian. Practitioners-anesthesiologists, as well as heads of departments, employees of departments, were invited to participate in the survey.

The survey results were imported into a Microsoft Excel spreadsheet for further analysis. Simple descriptive statistics were used for demographic data and numerical answers to individual questions. The answers, which included the free text were grouped by topic using simple qualitative techniques.

ELIGIBILITY:
Inclusion Criteria:

* experienced anesthesiologists

Exclusion Criteria:

* anesthesiologists out of practice

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Experienced anesthesiologists from most regions of Ukraine were interviewed.
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
The implication of the Helsinki Declaration on Patient Safety in the hospital | 2 months
  The implication of the Helsinki Declaration on Patient Safety in hospital

SECONDARY OUTCOMES:
The use of clinical protocols | 2 months
  The use of clinical protocols
Keeping records of anesthesia complications | 2 months
  Keeping records of anesthesia complications
The use of the WHO Safe Surgery checklist | 2 months
  The use of the WHO Safe Surgery checklist

CONTACTS AND LOCATIONS:
Overall Officials: Iurii Kuchyn, PhD, Study Director — Bogomolets National Medical University
Locations (1):
- Bogomolets NMU, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Staender SE, Mahajan RP. Anesthesia and patient safety: have we reached our limits? Curr Opin Anaesthesiol. 2011 Jun;24(3):349-53. doi: 10.1097/ACO.0b013e328344d90c. PMID 21330916
- [Background] Horton JB, Reece EM, Broughton G 2nd, Janis JE, Thornton JF, Rohrich RJ. Patient safety in the office-based setting. Plast Reconstr Surg. 2006 Apr;117(4):61e-80e. doi: 10.1097/01.prs.0000204796.65812.68. PMID 16582768
- [Background] Mellin-Olsen J, Staender S, Whitaker DK, Smith AF. The Helsinki Declaration on Patient Safety in Anaesthesiology. Eur J Anaesthesiol. 2010 Jul;27(7):592-7. doi: 10.1097/EJA.0b013e32833b1adf. PMID 20520556
- [Background] Balzer F, Spies C, Schaffartzik W, Pappert D, Wernecke KD, Kuhly R, Boemke W. Patient safety in anaesthesia: assessment of status quo in the Berlin-Brandenburg area, Germany. Eur J Anaesthesiol. 2011 Oct;28(10):749-52. doi: 10.1097/EJA.0b013e328348ee35. No abstract available. PMID 21785357
- [Background] Wu HHL, Lewis SR, Cikkelova M, Wacker J, Smith AF. Patient safety and the role of the Helsinki Declaration on Patient Safety in Anaesthesiology: A European survey. Eur J Anaesthesiol. 2019 Dec;36(12):946-954. doi: 10.1097/EJA.0000000000001043. PMID 31268913
- [Background] McColl E, Jacoby A, Thomas L, Soutter J, Bamford C, Steen N, Thomas R, Harvey E, Garratt A, Bond J. Design and use of questionnaires: a review of best practice applicable to surveys of health service staff and patients. Health Technol Assess. 2001;5(31):1-256. doi: 10.3310/hta5310. No abstract available. PMID 11809125
- [Background] Kelley K, Clark B, Brown V, Sitzia J. Good practice in the conduct and reporting of survey research. Int J Qual Health Care. 2003 Jun;15(3):261-6. doi: 10.1093/intqhc/mzg031. PMID 12803354
- [Derived] Bielka K, Kuchyn I, Semenko N, Kashchii U, Pliuta I. Patient safety during anesthesia in Ukraine: national audit results. BMC Anesthesiol. 2022 May 27;22(1):164. doi: 10.1186/s12871-022-01704-7. PMID 35624436